CLINICAL TRIAL: NCT07290634
Title: Comparative Outcomes of Prothrombin Complex Concentrate and Recombinant Activated Factor VIIa in Trauma-Associated Massive Transfusion: A Retrospective Cohort Study
Brief Title: Comparative Outcomes of PCC and Recombinant Activated Factor VIIa in Trauma-Associated Massive Transfusion
Status: Recruiting | Type: Observational
Sponsor: Zeliha Alicikus (Other Government)
Responsible Party: Sponsor-Investigator, Zeliha Alicikus, Head of Anesthesiology and Reanimation department,Assoc Prof, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Other Study IDs: AYTEN-2 FACTOR
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Thromboembolus; Massive Blood Transfusion; Thrombocytopenia; Trauma
MeSH Terms: conditions — Thromboembolism; Thrombocytopenia; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PCC group: patients receiving PCC during resuscitation
  Interventions: Procedure: Number of Participants with massive blood transfusion
- rFVIIa group: patients receiving rFVIIa
  Interventions: Procedure: Number of Participants with massive blood transfusion
- Combination group: patients receiving both PCC and rFVIIa
  Interventions: Procedure: Number of Participants with massive blood transfusion
- Control group: patients who received standard resuscitation without PCC or rFVIIa
  Interventions: Procedure: Number of Participants with massive blood transfusion

INTERVENTIONS:
Procedure: Number of Participants with massive blood transfusion — evaluate the impact of Prothrombin Complex, recombinant activated factor VII, and their combination on outcomes in adult trauma patients undergoing massive transfusion.

SUMMARY:
This study aims to compare the incidence of thromboembolic complications among trauma patients receiving PCC, rFVIIa, both agents, or neither during massive transfusion. Secondary objectives include comparing mortality, transfusion requirements, intensive care unit (ICU) and hospital length of stay, ventilator-free days, and the incidence of transfusion-associated adverse events such as transfusion-related acute lung injury (TRALI) and transfusion-associated circulatory overload (TACO). Subgroup analyses will evaluate outcomes in patients with and without laboratory-confirmed TIC (INR >1.2).

DETAILED DESCRIPTION:
Trauma-induced coagulopathy (TIC) is a multifactorial disorder that occurs in nearly one-third of severely injured patients and is closely linked to increased transfusion requirements, multiorgan failure, and higher mortality rates. Despite progress in trauma care and surgical interventions, hemorrhage and TIC remain leading contributors to preventable trauma-related deaths.

Conventional resuscitation approaches primarily involve fresh frozen plasma (FFP) and platelet transfusions; however, these blood products are constrained by delayed availability, large infusion volumes, and inconsistent concentrations of clotting factors. In addition, transfusing large amounts of plasma increases the risk of transfusion-associated circulatory overload (TACO) as well as transfusion related acute lung injeury (TRALI). By contrast, coagulation factor concentrates such as four-factor prothrombin complex concentrate (4F-PCC) and recombinant activated factor VII (rFVIIa) provide more rapid correction of deficiencies, require smaller infusion volumes, allow standardized dosing, and reduce logistical challenges.

Both randomized and observational investigations have explored the utility of PCC in TIC. The PROCOAG randomized clinical trial found no significant reduction in blood product use within 24 hours when PCC was given early compared with placebo, but reported a higher rate of thromboembolic complications . Mechanistic analyses demonstrated that PCC effectively enhanced thrombin generation, supporting its biological activity but also explaining the elevated thrombotic risk . A recent meta-analysis of randomized and cohort studies likewise showed that PCC reduced transfusion requirements but did not decrease mortality, while raising concerns over thromboembolic events at higher doses .

Systematic reviews published in recent years have drawn divergent conclusions. Some suggest that PCC may be most effective when used in carefully selected patients, often in conjunction with plasma, fibrinogen, or tranexamic acid. In contrast, Ovesen et al. highlighted that evidence from randomized trials remains insufficient to establish whether PCC is superior or inferior to other interventions in reducing clinically important outcomes or improving quality of life. Consequently, optimal dosing strategies and timing remain uncertain, and the balance between efficacy and thrombotic risk continues to be debated. As noted by Savi and Hawryluk , the absence of adequately powered clinical trials remains a major limitation for the development of standardized treatment algorithms. A recent qualitative synthesis incorporating seven observational studies and four randomized trials similarly concluded that the evidence base remains limited, underscoring the need for well-designed future research to clarify the role of PCC in TIC .

Recombinant activated factor VII, originally designed for patients with hemophilia and inhibitors, has also been employed off-label as a rescue therapy for uncontrollable bleeding in trauma. While initial studies indicated reductions in transfusion requirements, randomized trials failed to demonstrate a survival advantage and revealed higher thromboembolic risk, particularly in patients with preexisting cardiovascular disease . More recent systematic reviews confirm that although rFVIIa may achieve hemostasis in selected life-threatening cases, its routine use in unselected trauma patients is not supported .

Overall, available evidence suggests that both PCC and rFVIIa have the capacity to correct TIC, yet their safety profiles and impact on patient outcomes remain uncertain . Direct comparative research evaluating PCC, rFVIIa, and their potential combined use in real-world trauma practice is urgently needed to better define their influence on transfusion requirements, thrombotic events, and survival.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Trauma patients directly admitted from the scene with highest-level trauma activation: Injury -Severity Score (ISS) >15.
* Requirement for massive transfusion, defined as ≥3 units packed red blood cells (PRBC) within the first hour or ≥10 PRBC within the first 24 hours

Exclusion Criteria:

* Traumatic cardiac injury
* Death anticipated within the first hour of admission: ISS score >49
* Pre-injury anticoagulant therapy
* Known pregnancy
* Pre-injury terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a retrospective cohort study conducted between 1 January 2023 to 1 October 2025 at University of Florida Jacksonville trauma center. The study will evaluate the impact of Prothrombin Complex, recombinant activated factor VII, and their combination on outcomes in adult trauma patients undergoing massive transfusion.
Sampling Method: Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
thromboembolic events | 28 days
  Number of Participants with venous thrombosis, pulmonary embolism, ischemic stroke, mesenteric ischemia

SECONDARY OUTCOMES:
ICU and hospital stay | 28 days
  length of stay day

CONTACTS AND LOCATIONS:
Overall Officials: AYTEN SARAÇOĞLU, Prof,MD, Study Director — Florida University Jacksonville
Locations (1):
- UF Health Jacksonville (Shands Hospital), Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No